CLINICAL TRIAL: NCT00173680
Title: Methylation Status of CD44 Promoter Region in Primary Lung Cancer
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Other Study IDs: 9461700826
Record Dates: First submitted 2005-09-12; First posted 2005-09-15 (Estimated); Last update posted 2005-11-24 (Estimated); Status verified 2005-08

CONDITIONS: Non-Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Retrospective

SUMMARY:
This project is to study the methylation status of the transcriptional regulatory region of CD44 gene in surgically resected NSCLC specimens and normal lung tissue, correlate the methylation status of promoter region with the expression of CD44 gene, and analyze if methylation is associated with survival.

DETAILED DESCRIPTION:
CD44 is a cell surface receptor for the extracellular matrix hyaluronan. It mediates adhesion of cells to the extracellular matrix. Its ability to organize extracellular matrix into a medium is also used by cancer cells in their becoming metastatic. Invasive tumor cells are frequently observed to bind hyaluronate.

CD44 gene is made up of 20 exons, at least 10 of which are variably expressed due to alternative splicing of the mRNA. The standard form, CD44s, has a coding sequence of exons 1-5 and 16-20. Variant isoforms (CD44v), all larger, arise from alternative splicing of combinations of exons 6-15 (v1-10). A variant isoform CD44 can induce metastasis of a rat pancreatic carcinoma. Studies in human tumors, however, have produced variable results. Some breast cancers demonstrate positive correlation between CD44v expression and tumor progression, while others lack any correlation. Some colorectal tumors even show an inverse correlation. CD44 has also been demonstrated to be a metastasis suppressor gene for prostate cancer. Thus, CD44 may be a marker for metastasis for some tumors, but not for others, and it may actually be a metastasis suppressor gene for yet another groups of tumors.

For primary lung cancer, the correlation between CD44 expression and tumor metastasis has not been established. The metastasis-prone small cell lung cancer rarely showed any immunohistochemical staining for CD44s or CD44v. For non-small cell lung cancer (NSCLC), some studies showed positive correlation between immunohistochemical CD44v expression and tumor progression, while others showed no correlation. Our own study using RT-PCR, sequencing and immunohistochemical staining showed that in pulmonary adenocarcinoma, CD44v6 expression is down-regulated as the disease progressed. Based on our finding, and the observation that CD44s and CD44v expression are low in metastasis-prone small cell lung cancer, we assue that CD44 is a metastasis suppressor gene which is inactivated in lung cancers. Because in prostate cancer DNA hypermethylation has been shown to be related to the down-regulation of CD44 gene, we plan to study the methylation status of the transcriptional regulatory region of CD44 gene in primary lung cancer. We'll study CD44 expression by immunohistochemistry, the methylation status of CD44 regulatory region by sequencing of the bisulfite-modified genomic DNA, and correlate these two findings with each other, and with histologic type, tumor staging and survival.

ELIGIBILITY:
Inclusion Criteria:

* Non-small cell lung cancer

Exclusion Criteria:

* No

Min Age: 0 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40
Dates: Start 2005-08

CONTACTS AND LOCATIONS:
Overall Officials: LINA LEE, MD,PhD, Principal Investigator — Department of Labrotoary Medicine, National Taiwan University Hospital Taipei
Locations (1):
- Department of Laboratory Medicine, Nation Taiwan University Hospital, Taipei, Taiwan